CLINICAL TRIAL: NCT02396121
Title: Évaluation de l'évolution du Statut Nutritionnel en Micronutriment Chez Les Patients âgés dénutris bénéficiant d'Une complémentation Nutritionnelle Orale
Brief Title: Micronutrient and Malnourished Elderly
Acronym: Reboot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12.01.FR.NHS
Record Dates: First submitted 2015-02-04; First posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-02

CONDITIONS: Malnourished Elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interventional (Experimental): Administration of 1 bottle of an oral nutritional supplement, Renutryl® Booster (600 kcal), during 28 days.
  Interventions: Dietary Supplement: Oral nutritional supplement : Renutryl® Booster

INTERVENTIONS:
Dietary Supplement: Oral nutritional supplement : Renutryl® Booster

SUMMARY:
The purpose of this study is to evaluate the micronutrient status of malnourished elderly after oral nutritional supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Age : above or equal to 70 years

AND :

* Weight loss above or equal to 5% in one month
* OR weight loss above or equal to 10% in 6 months
* OR BMI between 18 and 21
* OR albuminaemia between 30 and 35 g/L
* OR MNA-SF less or equal to 7

Exclusion Criteria:

* Severe malnutrition
* Contraindication to oral nutrition
* Severe pathologies
* Inflammatory syndrome (CRP > 30 mg/L)
* Severe dementia (Mini Mental Score < 10)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 67 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in micronutrients status after 28 days | 28 days
  Biological analyses of micronutrient

SECONDARY OUTCOMES:
Nutritional status | 28 days
  Weight, albumin, transthyretin, CRP, Mini Nutritional Assessment Short-Form (MNA-SF)
Body composition | 28 days
  Impedance measurement
Compliance | 28 days
  Compliance measured by bottle weight before and after consumption
Autonomy | 28 fays
  "Get up and go" test